CLINICAL TRIAL: NCT06073704
Title: Effects of Antimicrobial Photodynamic Therapy in Non-surgical Periodontal Treatment of Patients with Obesity
Brief Title: Effects of Adjunct Antimicrobial Photodynamic Therapy in Periodontal Treatment of Patients with Obesity
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Carla Andreotti Damante, Associate professor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Obesity and Periodontitis
Record Dates: First submitted 2023-09-25; First posted 2023-10-10 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Periodontitis; Obesity
Keywords: periodontitis; obesity
MeSH Terms: conditions — Periodontitis; Obesity | interventions — Photochemotherapy; Tooth Exfoliation; Root Planing

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will be masked using a sham laser. Outcomes assessor will be blinded in relation to naming of the experimental groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Antimicrobial Photodynamic therapy adjunct to scaling and root planing (Experimental): Treatment of scaling and root planing followed by antimicrobial photodynamic therapy with methylene blue (100 micrograms/ml) and red laser
  Interventions: Procedure: antimicrobial photodynamic therapy (aPDT)
- Control (Active Comparator): Treatment of scaling and root planing.
  Interventions: Procedure: Control

INTERVENTIONS:
Procedure: antimicrobial photodynamic therapy (aPDT) — Scaling and root planing followed by antimicrobial photodynamic therapy
  Other Names: Photodynamic therapy; Photochemotherapy
  Arms: Antimicrobial Photodynamic therapy adjunct to scaling and root planing
Procedure: Control — Treatment of scaling and root planing
  Other Names: scaling and root planing
  Arms: Control

SUMMARY:
The goal of this clinical trial is to compare the effects of adjuvant antimicrobial photodynamic therapy (aPDT) as an adjuvant of scaling and root planing with scaling and root planing alone for periodontal treatment in patients with periodontal disease and obesity. The main question it aims to answer are: Does adjuvant aPDT improves periodontal health? Are there differences in the proteomic profile of gingival fluid after both treatments? Participants will receive scaling and root planing complemented or not by aPDT. Results will be collected after 1, 3, and 6 months. Researchers will compare adjuvant aPDT treatment to regular treatment to see if it promotes reduction in inflammation and improvement in periodontal health.

ELIGIBILITY:
Inclusion Criteria:

* Obesity (grade II and III classified according to Body Mass Index)
* Periodontitis stage II to IV
* Presence of at least 20 teeth excluding 3rd molars.

Exclusion Criteria:

* Smokers
* Alcohol or drugs consumption
* Kidney disorders
* Pregnancy or lactation
* Use of antibiotics at the last 30 days
* Use of drugs that alter periodontal structures as phenytoin or ciclosporin
* Periodontal treatment at the last 6 months

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-10-09 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Probing depth | Baseline, 1, 3 and 6 months
  Changes in probing depth measured from the gingival margin to the bottom of periodontal sulcus or periodontal pocket by a periodontal probe in millimeters.
Clinical attachment level | Baseline, 1, 3 and 6 months
  Changes in clinical attachment level measured from the cemento-enamel junction to the bottom of periodontal sulcus or periodontal pocket by a periodontal probe in millimeters.

SECONDARY OUTCOMES:
Changes on bleeding on probing | Baseline, 1,3,and 6 months
  Changes in percentage of sites with bleeding after probing. Six sites per tooth are examined and presence/absence of bleeding is recorded.
Differences in proteomics | baseline, 3 and 6 months
  Changes in inflammatory proteins after treatment by proteomics assay. Presence or absence of proteins in gingival fluid are compared before and after treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Bauru School of Dentistry, Bauru, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vohra F, Akram Z, Bukhari IA, Sheikh SA, Javed F. Short-term effects of adjunctive antimicrobial photodynamic therapy in obese patients with chronic periodontitis: A randomized controlled clinical trial. Photodiagnosis Photodyn Ther. 2018 Mar;21:10-15. doi: 10.1016/j.pdpdt.2017.10.022. Epub 2017 Oct 27. PMID 29111391
- [Background] da Silva-Junior PGB, Abreu LG, Costa FO, Cota LOM, Esteves-Lima RP. The effect of antimicrobial photodynamic therapy adjunct to non-surgical periodontal therapy on the treatment of periodontitis in individuals with type 2 diabetes mellitus: A systematic review and meta-analysis. Photodiagnosis Photodyn Ther. 2023 Jun;42:103573. doi: 10.1016/j.pdpdt.2023.103573. Epub 2023 Apr 14. PMID 37062511